CLINICAL TRIAL: NCT06248372
Title: The Investigation of the Effects of Attentional Focus Strategies on Pain, Disability, Posture, Quality of Life, and Depression in Patients With Myofascial Pain Syndrome
Brief Title: Attentional Focus Strategies in Exercise in Patients With Myofascial Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yeditepe University (Other)
Responsible Party: Principal Investigator, Yagmur Barlas, Master Degree Student, Yeditepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Yagmur
Record Dates: First submitted 2024-01-23; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Myofascial Pain Syndrome
Keywords: Pain; Pressure Pain Threshold; Quality of Life; Depression; Posture; Myofascial Pain Syndrome; Attentional Focus Strategies
MeSH Terms: conditions — Myofascial Pain Syndromes; Pain; Depression | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- External Focus Group (EFG) (Experimental): Receive exercise program that includes strengthening and stretching exercises however this group will focus on environmental cues apart from body movement by using metaphors or analogies.
  Interventions: Other: Exercise
- Internal Focused Group (IFG) (Experimental): Receive exercise program that includes strengthening and stretching exercises however this group will follow internal cues directing attention to the body movement (i.e., joint movement) while doing exercises.
  Interventions: Other: Exercise
- Control Group (CG) (Other): Receive exercise program that includes strengthening and stretching exercises however, this group will not focus on any attentional cues while doing exercises.
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Both groups will receive the same exercise program that includes strengthening and stretching exercises except for the verbal instructions which shift attention to the internal or external environment or no attentional instructions for the control group.

SUMMARY:
Attentional focus is a concept of motor learning and the usage of this concept promotes exercise-induced muscular adaptations and affects motor performances. In practice,two main verbal instructions are directing the focus of attention; external focus (EFA) and internal focus of attention (IFA). Several studies show the results related with different health conditions. However, there is not enough studies to investigate the effectiveness of these attentional focus strategies in exercise regimes in patients with musculoskeletal problem. Thus, the study will be the first to investigate the effectiveness of attentional focus strategies in patients with neck and upper back myofascial pain syndrome (MPS) which is the most common syndrome of musculoskeletal problems.

DETAILED DESCRIPTION:
When investigating the literature studies, there is insufficient evidence to determine which attentional focus strategies are more effective for improving function and decreasing pain in different health conditions. In most of the studies duration of symptoms of patients was not mentioned and there are no studies that directly compare EFA and IFA and report the effects on pain or functional outcomes in musculoskeletal conditions.Additionally, one study investigated the effectiveness of attentional focus strategies used in a training program but not in a musculoskeletal problem.

Thus, the study aims to investigate the effectiveness of attentional focus strategies in patients with neck and upper back MPS in terms of pain, pressure pain threshold, quality of life, depression, disability, and posture parameters.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic MPS in the neck and upper back region (upper and middle trapezius, levator scapulae, rhomboids, infraspinatus, and supraspinatus muscles) confirmed by a physician,
* Pain lasting more than 3 months with a pain intensity is 3 or higher according to numeric pain rating scale (NPRS⩾3).

Exclusion Criteria:

* Fibromyalgia syndrome, cervical disc pathologies, malignancy, neurologic and/or inflammatory diseases, history of neck, shoulder, upper back surgery and trauma, other medical conditions that limit participation in exercise.
* Pregnancy
* Individuals being involved in physiotherapy or exercise sessions for at least 4 weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-01-30 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | through study completion;an average 8 months
  It is a common scale to measure the perceived level of pain intensity on a numeric scale that usually includes 11 numbers. The participant is instructed to select the number that best reflects the intensity of pain experienced, with 0 representing one extreme of pain (e.g., no pain) and 10 representing the other extreme (e.g., pain as bad as it could be).
Pressure Pain Threshold (PPT) | through study completion;an average 8 months
  A digital algometer (Jtech Medical Commander Echo) will be applied to measure the pressure pain threshold of the four most painful myofascial trigger points on both sides of the upper and middle trapezius, levator scapulae, rhomboids, infraspinatus, and supraspinatus. It has a circular flat tip of 1 cm2 which will be pushed slowly to the skin over the trigger points after exploration of a taut band with a normalized speed until the subject presses a switch when the compression sensation alters to pain. This process will repeat three times with a 30-second rest in between and their average will be considered as pressure pain threshold.

SECONDARY OUTCOMES:
New York Posture Rating Chart (NPRC) | through study completion;an average 8 months
  In this rating chart, posture changes that may occur in 13 different parts of the body are monitored and scored. Accordingly, 5 points will be given if the person's posture is correct, 3 points will be given if the person's posture is moderately impaired, and 1 point will be given if the person's posture is seriously impaired. The total score obtained as a result of the test. 65 is the maximum score while the minimum score is 13.
Neck Disability Index (NDI) | through study completion;an average 8 months
  It is a self-report questionnaire used to determine how neck pain affects a patient's daily life and to assess the self-rated disability of patients with neck pain. Each section is scored on a 0 to 5 rating scale, in which 0 means 'no pain' and 5 means 'worst imaginable pain'. The lower score means the individual's daily living activities are affected less.
Beck Depression Inventory (BDI) | through study completion;an average 8 months
  It is a 21-question inventory for measuring the severity of depression. Each question has a set of four possible responses scored between 0 to 3. A total score shows the severity of depression. 0- 9 indicates minimal depression,10-18: indicates mild depression,19-29: indicates moderate depression, and 30-63: indicates severe depression. Higher total scores indicate more severe depression the individual has.
SF-12 Questionnaire (SF-12) | through study completion;an average 8 months
  It is a self-reported outcome measure assessing the impact of health on an individual's everyday life. It is generally used to measure the quality of life of individuals. SF-12 is a short form of SF-36 by taking 12 different items. There are two components which is physical and mental. A higher score indicates good health status.

IPD SHARING:
Plan to Share IPD: Undecided